CLINICAL TRIAL: NCT01605643
Title: Biomarker Feedback to Motivate Tobacco Cessation in Pregnant Alaska Native Women: Phase 1
Brief Title: Biomarker Feedback to Motivate Tobacco Cessation in Pregnant Alaska Native Women
Acronym: MAW
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Alaska Native Tribal Health Consortium (Other); University of California, San Francisco (Other); University of Minnesota (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christi Patten, Professor of Psychology, Mayo Clinic
Other Study IDs: 11-001144; U54CA153605 (NIH)
Record Dates: First submitted 2012-05-07; First posted 2012-05-25 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Cancer; Tobacco Use; Pregnancy
Keywords: cancer; tobacco use; pregnancy
MeSH Terms: conditions — Neoplasms; Tobacco Use

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — urine and serum specimen samples collected from mother and infant pairs
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Use of tobacco is very high among Alaska Native women. The investigators are conducting a three phase study. The first phase will examine biomarkers of tobacco exposure in pregnant women and their newborns. The second phase is a qualitative study to translate the biomarker findings into intervention messages. The third phase is a pilot of the biomarker feedback intervention compared with a control condition.

DETAILED DESCRIPTION:
Developing effective tobacco cessation interventions during pregnancy for American Indian and Alaska Native people is a national priority and will contribute to the U.S. public health objective of reducing tobacco-related cancer health disparities. The proposed project builds on our successful partnership with the Alaska Native community and previous work with Alaska Native pregnant women. We propose to develop and test a novel biomarker feedback intervention relating cotinine levels in the urine of pregnant women with the woman and infant's likely exposure to the tobacco specific nitrosamine and carcinogen 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone) (NNK). This 5-year project will be conducted in three phases. In Phase 1 we will utilize a non-randomized, clinical observational trial to examine biomarkers of nicotine and carcinogen exposure (urine cotinine and total NNAL [a metabolite of NNK], respectively) among 150 maternal-infant pairs with assessments conducted during pregnancy and at delivery. In Phase 2, we will obtain qualitative feedback on the findings from Phase 1 through individual interviews conducted with 32 women who use tobacco to develop the biomarker feedback intervention messages. Phase 3 will consist of a formative evaluation of the biomarker feedback intervention with 80 pregnant women using a two-group randomized design to assess the intervention's feasibility and acceptability, and the biochemically confirmed abstinence rate at the end of pregnancy. All phases of the project will be guided by a Community Advisory Committee. Each phase is an important step to advance our understanding of the potential for biomarker feedback as a strategy to help Alaska Native pregnant women quit tobacco use. The potential reach of the intervention is significant from a public health perspective as over 600 tobacco users deliver each year at the Alaska Native Medical Center in Anchorage where the proposed project will take place. Developing effective interventions for tobacco cessation during pregnancy is important to reduce adverse health consequences for the mother and neonate and future risk of tobacco-caused cancers.

ELIGIBILITY:
Inclusion Criteria:

To be eligible the woman must:

1. be Alaska Native,
2. be aged 18 years or older,
3. provide written informed consent,
4. be currently pregnant (1st, 2nd or 3rd trimester), and
5. plan to deliver at the ANMC. An additional inclusion criterion for current tobacco users is any use in the past 7 days. Our preliminary studies indicate that women may use more than one form of tobacco. To enhance feasibility of recruitment and generalizability, women will not be excluded if they use more than one form of tobacco. Instead, group composition will be based on the primary type of tobacco used. An additional inclusion criterion for non-tobacco users is no use of any form of tobacco in the last 6 months.

Exclusion Criteria:

1. Women will be excluded if they have used nicotine replacement therapy (NRT) or have participated in a behavioral or pharmacological tobacco cessation program within the past 30 days.
2. Alcohol and other drug use will not be an exclusionary criterion because the biomarkers are specific to tobacco exposure.

Max Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pregnant women will be recruited through prenatal care
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
NNAL | delivery

SECONDARY OUTCOMES:
cotinine | participants will be followed during pregnancy until approximately week 40 gestation and Infants will be assessed at birth only
  tobacco exposure measured during pregnancy and at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Christi A Patten, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Alaska Native Tribal Health Consortium, Anchorage, Alaska, United States